CLINICAL TRIAL: NCT04369248
Title: Hepassocin Levels in Patients With Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Fatma ketenci gencer (Other Government)
Responsible Party: Sponsor-Investigator, Fatma ketenci gencer, principal invastigator, Gaziosmanpasa Research and Education Hospital
Organization: Gaziosmanpasa Research and Education Hospital (Other Government)
Other Study IDs: GaziosmanpasaTREH19
Record Dates: First submitted 2020-04-26; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Hepassocin (Hepatocyte-derived Fibrinogen-related Protein 1); Polycystic Ovary Syndrome; Obesity; Insulin Resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Early follicular phase day 3 in case of menstruating and random day for amenorrheic patients was chosen for blood sampling after 8 hour of fasting. The blood samples were obtained from the antecubital vein via a vacutainer. Process of samples was achieved within maximum 1 hour and serum sample was stored in -80 for hepassocin work-up after 5 minutes of centrifuge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: 30 healthy women with BMI < 30 between 18 and 35 years old
  Interventions: Other: hepassocin
- Non-obese PCOS: 2003 Rotterdam ESHRE/ASRM PCOS Consensus Criteria were used to diagnose PCOS that fulfilled at least two of the followings: chronic oligo-anovulation, clinic or biochemical hyperandrogenism and presence of polycyctic ovary by ultrasound (Rotterdam). Oligo-anovulation is defined as periods lasting more than 35 days and/or amenorrhea. Clinic or biochemical hyperandrogenism is defined as the presence of acnes and/ or Ferriman-Galleway modified score >8 and/ or hyperandrogenemia defining the testosterone level > 0.6 ng/ml (2 nmol/l) and/or dehydroepiandrosterone level > 3 ng/ml (10.5 nmol/l). Polycyctic ovaries are defined as the presence of more than 12 follicules 2-9 mm in diameters or ovarian volume >10 cm3 under transvaginal or abdominal ultrasound. non-obese group are the women BMI < 30 between age of 18 and 35.
  Interventions: Other: hepassocin
- Obese PCOS: Obese group are the women with BMI > 30 between age of 18 and 35.
  Interventions: Other: hepassocin

INTERVENTIONS:
Other: hepassocin — hepassocin levels in polycystic ovary syndrome

SUMMARY:
The investigators aimed to investigate hepassocin levels in patients with polycystic ovary syndrome (PCOS). There are 3 groups aged between 18 and 35 years as non-obese healthy women, non-obese women with PCOS, and obese women (BMI>30) with PCOS.

DETAILED DESCRIPTION:
Hepassocin, also known as Fibrinogen-like-protein or hepatocyte-derived fibrinogen-related protein 1, is a new marker for obesity and insulin resistance. In hepatic injury, it protects liver cells and promotes regeneration. High levels of hepassocin was shown to be independently associated with HOMA-IR and diabetes. Since insulin resistance is known to be seen in patients with PCOS, it may be expected that hepassocin levels may be higher in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* 60 patients with PCOS aged between 18 and 35 and age-matched 30 healthy women with BMI<30

Exclusion Criteria:

Premature ovarian failure (FSH >30 mIU/mL), tumors secreting androgens, non-classical congenital adrenal hyperplasia, Cushing syndrome and irregular menses due to thyroid dysfunction (TSH >5 mIU/L ), hyperprolactinemia, more than twofold high transaminase levels (>70 U/L), patients with cigarette smoking, alcohol consumption, oral contraceptives use, medications that are affecting liver function test, insulin metabolism and lipid metabolism, patients with a history of chronic diseases such as diabetes mellitus, hypertension, chronic liver disease, chronic kidney disease, autoimmune disease, inflammatory disease, malignant disease, bleeding disorders, and thrombosis were also excluded. All the patients were beta-HCG, hepatitis B surface antigen, and hepatitis C antibody negative.

-

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 60 patients with PCOS aged between 18 and 35 and age matched 30 healthy women with BMI < 30 were enrolled to the study.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Hepassocin levels in patients with polycystic ovary syndrome | January 2020-March 2020
  hepassocin levels should be increased in polycyctic ovary syndrome due to its relation with insulin resistance.

CONTACTS AND LOCATIONS:
Overall Officials: fatma ketenci gencer, Study Director — Gaziosmanpasa Taksim Education and Research Hospital; sibel bektas, Study Chair — Gaziosmanpasa Taksim Education and Research Hospital
Locations (1):
- Gaziosmanpasa Taksim Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided